CLINICAL TRIAL: NCT05797493
Title: Panomic Approach to Immune-Connected Assays in Small Cell Lung Cancer
Acronym: PICASSO
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Bria Emilio, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 5061
Record Dates: First submitted 2023-03-16; First posted 2023-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Small Cell Lung Cancer
Keywords: sclc; immunotherapy
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — atezolizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ES-SCLC: ES-SCLC receiving upfront chemo-immunotherapy
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Atezolizumab — Upfront chemo-immunotherapy

SUMMARY:
The scope of the PICASSO project is to apply an innovative patient-based pan-omic approach to immune-assays, that will include multi-omics tumour characterization (genome, proteome, transcriptome), blood immune-cells and cytokine profiling, serological screening for paraneoplastic autoantibodies, clinical and metabolic measurements.

The PICASSO project is aimed to validate in real world population the predictive role of SCLC transcriptomic classification (particularly, I-SCLC subtype) and to explore correlations with dynamic changes in peripheral blood immunity. Additionally, investigators expected to validate the predictive/prognostic role of emerging new variables, including metabolic-induced meta-inflammation alterations and subclinical auto-immunity.

ELIGIBILITY:
Inclusion Criteria:

1. histologically- or cytologically-documented extensive-stage SCLC
2. to have received upfront treatment with Cisplatin/Carboplatin, etoposide and anti PD1/PD-L1 inhibitors
3. No evidence of brain metastases at diagnosis
4. ECOG PS 0-2
5. adult patients (aged ≥ 18 years) at diagnosis;
6. signing of informed consent approved by the local Ethic Committee

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ES SCLC patients treated with first line chemo-immunotherapy (EP-IO
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-10-04 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
PFS | Up to 60 months
  Time from treatment start until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
OS | Up to 60 months
  Time from treatment start to the date of death from any cause, assessed up to 60 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: No